CLINICAL TRIAL: NCT06041646
Title: Characterization of Tachyphylaxis, Tolerance, and Withdrawal After Discontinuation of Igalmi in Frequently Agitated Schizophrenic or Bipolar Patients After 7 Days of PRN Treatment
Brief Title: Tachyphylaxis, Tolerance, & Withdrawal Post Treatment With Igalmi for Agitation in Schizophrenia or Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: BioXcel Therapeutics Inc (Industry)
Collaborators: Lotus Clinical Research, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BXCL501-404
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Results first posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Bipolar Disorder; Schizophrenia; Agitation,Psychomotor; Schizo Affective Disorder; Schizophreniform Disorders
Keywords: Agitation; Schizophrenia; Bipolar; Dexmedetomidine; tachyphylaxis; tolerance; withdrawal; PRN treatment; Open-Label; PEC; CGI; ACES; Safety; Tolerability; Igalmi
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia; Psychomotor Agitation; Psychotic Disorders | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Open-Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active Treatment - 180 mcg of Igalmi (dexmedetomidine) (Other): An initial dose of 180 µg of Igalmi as needed for the treatment of agitation over a period of 7 days. In the event of persistent or recurrent agitation, investigators may choose to repeat dose at 90 μg after the 2-hour time point in the absence of dose-limiting adverse events or safety concerns. A maximum of 2 repeat doses will be allowed in a 24-hour period.
  Interventions: Drug: Sublingual film containing Igalmi

INTERVENTIONS:
Drug: Sublingual film containing Igalmi — Sublingual film containing 180 µg of Igalmi (dexmedetomidine)
  Other Names: Dexmedetomidine; BXCL501

SUMMARY:
This is an in-clinic, single arm, open-label study assessing tachyphylaxis, tolerance, and withdrawal following repeated doses of Igalmi in adult males and females with agitation associated with schizophrenia or bipolar disorder.

DETAILED DESCRIPTION:
This is an in-clinic, single arm, open-label study assessing tachyphylaxis, tolerance, and withdrawal following repeated doses of Igalmi in adult males and females (18 to 65 years old, inclusive) with agitation associated with schizophrenia or bipolar disorder. Subjects will be screened for eligibility within 15 days of first dose and no study procedures will occur unless subjects provide written informed consent. Subjects will receive single doses of 180 μg of Igalmi as needed for the treatment of agitation over a period of 7 days followed by a 3- day follow-up period during which time no Igalmi will be administered in an effort to characterize any potential withdrawal. Subjects will sublingually self-administer Igalmi for an agitation episode that reaches a pre-dose PEC total score of 14 or greater, as determined by a trained rater. Safety assessments will be conducted before and after each dose. If the subject's agitation is recurrent or persistent, repeat doses of 90 µg may be administered (no more than 2 repeat doses within a 24-hour period) in the absence of any safety concerns or adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between the ages of 18 to 65 years, inclusive.
2. Subjects who have met DSM-5 criteria for schizophrenia, schizoaffective, or schizophreniform disorder or bipolar I or II disorder.
3. Subjects who are currently moderate to severely agitated at least 3 days a week.
4. Subjects who read, understand, and provide written informed consent.
5. Subjects who are in good general health prior to study participation as determined by a detailed medical history and in the opinion of the Principal Investigator.
6. Subjects who agree to use a medically acceptable and effective birth control method
7. Subjects must be willing to remain in-clinic for the duration of the study.

Exclusion Criteria:

1. Subjects with agitation caused by acute intoxication, including positive identification of alcohol by breathalyzer or drugs of abuse during screening.
2. Use of benzodiazepines or other hypnotics or antipsychotic drugs in the 6 hours before study treatment.
3. Subjects with congenital prolonged QT syndrome.
4. Prior treatment with Igalmi

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Risinger, MD, Study Chair — BioXcel Therapeutics
Locations (2):
- United States (2):
  - BioXcel Clinical Research Site, Little Rock, Arkansas
  - BioXcel Clinical Research Site, Rogers, Arkansas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in the United States from 02Oct2023 to 29Apr2024.
Period: Overall Study
Arm/Group | Active Treatment - 180 mcg of Igalmi (Dexmedetomidine)
Started | 29
Completed | 28
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Active Treatment - 180 mcg of Igalmi (Dexmedetomidine)
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (8.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 15
  More than one race | 1
  Unknown or Not Reported | 0
Diagnosis [Count of Participants; unit: Participants]
  Bipolar 1 or 2 | 17
  Schizophrenia | 10
  Schizoaffective disorder | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Positive and Negative Syndrome Scale- Excited Component (PEC) Total Score
Description: The Positive and Negative Syndrome Scale-Excited Component (PEC) includes 5 items-poor impulse control, tension, hostility, uncooperativeness, and excitement-each of which is rated from 1 (minimum) to 7 (maximum); the sum of these 5 items, the PEC total score, ranges from 5 (absence of agitation) to 35 (extremely severe).
Time Frame: Baseline and 2 hours post-dose for all doses administered over 7 days.
Population: For each dose the population consists only of patients who took that dose.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Treatment - 180 mcg of Igalmi (Dexmedetomidine)
Number analyzed (Participants) | 28
score on a scale
  Dose 1 | -10.4 (2.94)
  Dose 2: number analyzed (Participants) | 23
  Dose 2 | -10.0 (3.54)
  Dose 3: number analyzed (Participants) | 14
  Dose 3 | -10.1 (3.60)
  Dose 4: number analyzed (Participants) | 8
  Dose 4 | -9.8 (2.55)
  Dose 5: number analyzed (Participants) | 6
  Dose 5 | -11.5 (4.51)
  Dose 6: number analyzed (Participants) | 3
  Dose 6 | -8.7 (3.79)
  Dose 7: number analyzed (Participants) | 1
  Dose 7 | -11.0 (NA) — Not available as only one patient is included.

2. Primary Outcome: Clinical Global Impression - Improvement (CGI-I)
Description: The Clinical Global Impression - Improvement (CGI-I) for agitation in response to treatment measures the current level of agitation relative to the level of agitation prior to administration of study intervention. The CGI-I scores range from 1 to 7 with a score of 1 indicating very much improved, and a score of 7 indicating very much worse.
Time Frame: 2 hours post-dose for all doses administered over 7 days.
Population: For each dose only the patients who took that dose are included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Treatment - 180 mcg of Igalmi (Dexmedetomidine)
Number analyzed (Participants) | 28
score on a scale
  Dose 1 | 1.2 (0.50)
  Dose 2: number analyzed (Participants) | 23
  Dose 2 | 1.2 (0.39)
  Dose 3: number analyzed (Participants) | 14
  Dose 3 | 1.3 (0.47)
  Dose 4: number analyzed (Participants) | 8
  Dose 4 | 1.0 (0.00)
  Dose 5: number analyzed (Participants) | 6
  Dose 5 | 1.2 (0.41)
  Dose 6: number analyzed (Participants) | 3
  Dose 6 | 1.3 (0.58)
  Dose 7: number analyzed (Participants) | 1
  Dose 7 | 2.0 (NA) — Only one patient.

3. Secondary Outcome: Number of Participants With Adverse Events During the Follow-up Period
Description: Evaluation of withdrawal phenomenon based on the occurrence of adverse events such as tachycardia, systolic hypertension, nausea, or vomiting and the emergence of any new adverse events on ≥2 consecutive days of the 3-day off-treatment follow-up period.
Time Frame: Day 8 through Day 10
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment - 180 mcg of Igalmi (Dexmedetomidine)
Number analyzed (Participants) | 28
Participants | 0

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | Active Treatment - 180 mcg of Igalmi (Dexmedetomidine)
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 14/28
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment - 180 mcg of Igalmi (Dexmedetomidine) (N=28)
Headache (Nervous system disorders) | 3 (3)
Somnolence (Nervous system disorders) | 3 (4)
Dizziness (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 3 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Hypoesthesia oral (Gastrointestinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysmenorrhea (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/46/NCT06041646/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT06041646/SAP_001.pdf